CLINICAL TRIAL: NCT04907617
Title: The Effect of Active Warming During General Anaesthesia on Postoperative Body Temperature, Shivering, Thermal Comfort, Pain, Nausea and Vomiting in Adult Patients: A Randomised Controlled Trial Protocol
Brief Title: The Effect of Active Warming During General Anaesthesia on Postoperative Body Temperature, Shivering and Thermal Comfort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ozlem Sahin Akboga, Principal İnvestigator, Bozok University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: marmarabozok
Record Dates: First submitted 2021-05-22; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Nursing Caries; Postoperative Pain; Postoperative Nausea and Vomiting
Keywords: Perioperative Nursing; Body Temperature; Hypothermia; Shivering; Pain; Postoperative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Hypothermia; Pain

STUDY DESIGN:
Intervention Model Description: The participants in the study will be allocated to one of four groups. In the trial, the participants will be assigned to the interventions and registered by the first author of this study.After the induction of anaesthesia, forced-air warming as well as warmed IV and irrigation fluids will be applied to the first group, the second group will be heated with only forced-air warming device, the third group will receive only warmed IV and irrigation fluids, and the fourth group will be the control group without any intervention.
Who Masked: Participant
Masking Description: The participants will be blinded to the trial hypothesis and design to avoid being affected by the warming intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G1 (Experimental): After the induction of anaesthesia, the first group will be heated with only forced-air warming device.
  Interventions: Other: FAW
- G2 (Experimental): After the induction of anaesthesia, the second group will receive only warmed IV and irrigation fluids.
  Interventions: Other: Warmed fluids
- G3 (Experimental): After the induction of anaesthesia, forced-air warming as well as warmed IV and irrigation fluids will be applied to the third group
  Interventions: Other: Combination
- G4 (Experimental): After the induction of anaesthesia, the fourth group will be the control group without any intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: FAW — After the induction of anaesthesia, for patients assigned to groups 1 and 3, the cover of the forced-air warming device (Bair HuggerTM Warming Unit, Model 505, Augustine Medical Inc., Eden Prairie, MN, USA) will be covered over the patient, with the surgical site exposed, and the temperature adjustment of the device will be set to the maximum (43°C). Then, the temperature will be adjusted to maintain a patient temperature of at least 36.5°C. When the patient's body temperature reaches 37°C, the device will be turned off and it will be restarted at a temperature measurement of <36.5°C.
  Arms: G1
Other: Warmed fluids — In patients assigned to groups 2 and 3, intraoperative IV (Automer blood/fluid warming system, Acemedikal, South Korea) and irrigation fluids (Enthermic Warming Cabinet 1002W, Poland) will be given by heating to 37°C in a thermostatically controlled heating cabinet.
  Arms: G2
Other: Combination — After the induction of anaesthesia, for patients assigned to groups 3, the cover of the forced-air warming device (Bair HuggerTM Warming Unit, Model 505, Augustine Medical Inc., Eden Prairie, MN, USA) will be covered over the patient, with the surgical site exposed, and the temperature adjustment of the device will be set to the maximum (43°C). Then, the temperature will be adjusted to maintain a patient temperature of at least 36.5°C. When the patient's body temperature reaches 37°C, the device will be turned off and it will be restarted at a temperature measurement of <36.5°C.
  In patients assigned to groups 3, intraoperative IV (Automer blood/fluid warming system, Acemedikal, South Korea) and irrigation fluids (Enthermic Warming Cabinet 1002W, Poland) will be given by heating to 37°C in a thermostatically controlled heating cabinet.
  Arms: G3
Other: Control — The patients assigned to group 4 will only receive 'routine care'. They will not be given intraoperative forced-air warming or heated IV and irrigation fluids.
  Arms: G4

SUMMARY:
Adult patients who undergo surgery under general anaesthesia often experience inadvertent perioperative hypothermia. This common problem has serious consequences such as surgical site infection, coagulopathy, increased need for transfusion, altered drug metabolism and adverse cardiac events. Perioperative guidelines recommend warming the patient with a forced-air warming device and administering warmed intravenous and irrigation fluids to prevent intraoperative hypothermia. This study aims to investigate the effects of individual and combined use of intraoperative forced-air warming and warmed intravenous and irrigation fluids on postoperative body temperature, shivering, thermal comfort, pain, nausea and vomiting in adult patients receiving general anaesthesia.

DETAILED DESCRIPTION:
Background: Adult patients who undergo surgery under general anaesthesia often experience inadvertent perioperative hypothermia. This common problem has serious consequences such as surgical site infection, coagulopathy, increased need for transfusion, altered drug metabolism and adverse cardiac events. Perioperative guidelines recommend warming the patient with a forced-air warming device and administering warmed intravenous and irrigation fluids to prevent intraoperative hypothermia.

Objective: This study aims to investigate the effects of individual and combined use of intraoperative forced-air warming and warmed intravenous and irrigation fluids on postoperative body temperature, shivering, thermal comfort, pain, nausea and vomiting in adult patients receiving general anaesthesia.

Design and setting: This is a single centre randomised controlled clinical trial. A 2 x 2 factorial design will used in the experiment. Eligible patients will be randomly assigned to one of four groups.

Methods: After the induction of anaesthesia, forced-air warming as well as warmed intravenous (IV) and irrigation fluids will be applied to the first group, the second group will be warmed with only forced-air warming device, the third group will receive only warmed intravenous and irrigation fluids, and the fourth group will consist of the control group without any intervention. Blood and blood products to be applied intraoperatively to all groups will be heated to 37°C. The primary outcome measures are postoperative body temperature, shivering, thermal comfort, pain, nausea and vomiting. The primary results will be subjected to a two-way analysis of variance for covariants such as ambient temperature and volume of intraoperative fluids.

Participants: The trial will include patients aged ≥18 years who underwent surgery under general anaesthesia, whose duration of surgery was >1 hour, who belong to the class of American Society of Anesthesiologists I-III, who do not have any disability that would make communication difficult, and who provide written informed consent to participate in the study.

Discussion: The trial is designed to validate the effectiveness of these two interventions administered alone and in combination in maintaining perioperative normothermia and to assess whether they translate into improved patient outcomes.

* This trial is being carried out as Marmara University Institute of Health Sciences Doctorate Thesis in Nursing.

Funding: No funding

ELIGIBILITY:
Inclusion Criteria:

Being over the age of 18 Receiving general anesthesia, surgery time ≥ 1 hour in the American Society of Anesthesiologists (ASA) I-III class Not having any obstacle to make communication difficult İnformed written consent to participate in the study.

Exclusion Criteria:

Having surgery with local anesthesia Preoperative body temperature ≥38 0C or <36 0C Unapplied therapeutic hypothermia during the operation, Systemic infection in the patient, Mental retardation, Serious head injury, Brain damage disruption in temperature regulation, Taking medication to affect thermoregulation Unapplied IV fluids up to one hour before anesthesia induction.

Exclusion criteria is exitus and worsening for any reason in the general condition during and after the surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-09-18 (Estimated); Study Completion 2021-12-18 (Estimated)

PRIMARY OUTCOMES:
Body temperature | two days
  In the trial, the body temperature of the participants will be measured with a tympanic thermometer (Braun ThermoScan® 3, IRT 3030, Mexico, USA).
Thermal comfort scale | two days
  The thermal comfort of the patients will be measured with a 100-point thermal comfort scale based on self-reporting. The patients will be asked to score how comfortable they are with their body temperature [0 = extremities too cold; 50 = no discomfort (shivering or sweating); 100 = extremities too hot] on a scale of 0-100 points (Cobb et al., 2016). This numerical rating scale has been used effectively in previous studies on thermal comfort
Shivering | two days
  Shivering will be assessed using a 4-point bedside shivering assessment scale developed by Badjatia et al. (2008) [0 = no shivering; 1 = mild (shivering localised in the neck/thorax, only visible as an artefact on EEG or can be noted on palpation); 2 = moderate (intermittent shivering in the upper extremities ± thorax); 3 = severe (diffuse shivering or continuous shivering in the upper/lower extremities)]
Postoperative pain | two days
  The postoperative pain of the patients will be assessed with the Numerical Rating Scale (NRS) based on self-reporting. The obtained NRS score will be considered as 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain (Chou et al., 2016; Van Dijk et al., 2012).
Postoperative nausea and vomiting | two
  Based on a previous study, the presence of postoperative nausea and vomiting of the patients in the trial will be considered as follows: 0 = no nausea; 1 = nausea without vomiting; 2 = nausea with vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not suitable for making individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Sahin Akboga O, Gurkan A. Effects of Active Heating Methods on Body Temperature, Shivering, Thermal Comfort, Pain, Nausea and Vomiting During General Anesthesia: A Randomized Controlled Trial. Ther Hypothermia Temp Manag. 2024 Dec;14(4):269-281. doi: 10.1089/ther.2023.0049. Epub 2023 Nov 24. PMID 38011688